CLINICAL TRIAL: NCT03233633
Title: Marijuana in Combination With Opioids for Pain and Symptom Control in Hospice Patients
Brief Title: Marijuana in Combination With Opioids in Palliative and Hospice Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Connecticut Hospice Inc. (Other)
Responsible Party: Principal Investigator, Theodore Zanker MD, Principal Investigator, The Connecticut Hospice Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: WIRB Protocol 20161880-1167645
Record Dates: First submitted 2017-07-26; First posted 2017-07-28 (Actual); Results first posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Pain
Keywords: pain management; terminally ill
MeSH Terms: conditions — Pain; Agnosia | interventions — Medical Marijuana; Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single treatment arm (Other): marijuana adjuvant treatment group utilizing scheduled opioid therapy in inpatient hospice hospital setting
  Interventions: Drug: Medical Marijuana

INTERVENTIONS:
Drug: Medical Marijuana — oral capsule, high ratio CBD:THC
  Other Names: cannabidiol; medical cannabis

SUMMARY:
Study Objectives: Primary reduction of pain and reduction in overall opioid utilization. Secondary improvement in overall patient well being, weight stabilization with increased appetite, improved oxygen saturation, improvement or prevention of nausea and vomiting.

Study Rationale: To determine optimum use and dosing of medical marijuana (CBD:THC) for pain and symptom management.

Study Population: This study specifically will enroll cancer and non-cancer patients as a primary diagnosis suffering from pain and having a terminal illness (defined as having less than 6 months to live) requiring end of life care.

DETAILED DESCRIPTION:
Primary Endpoint: Primary reduction of pain and reduction in overall opioid utilization as evidenced by overall reduction in numeric pain scores and MME (Morphine Milliequivalents)

Secondary and Exploratory endpoints:Secondary improvement in overall patient well being, weight stabilization with increased appetite, improved oxygen saturation, improvement or prevention of nausea and vomiting. Endpoints evaluation will be based on change from Baseline using the Modified Edmonton Assessment Scale.

Study design: This will be an open-label study. Patients will choose to participate in a Marijuana adjuvant treatment group, receiving marijuana in combination with standard opioid therapy.

Subject number: Minimum 66 patients

Treatment Duration: Minimum 5 days

Duration of follow up: Patients' initial opioid dose, dosing schedule and numeric pain score will be recorded. For the duration of the study (at least five days) changes in opioid doses and numeric pain scores will be tracked daily.

Marijuana will be administered to the patient via oral route three times daily for at least five days. Patients will receive standardized CBD:THC product provided by NIDA.

On admission to the study, a modified Edmonton Symptom assessment scale to quantify baseline appetite, depression, nausea, vomiting, overall well-being, and anxiety.

Data Tracking: Primary objective tracking will include average numeric pain scores and number of opioid dosage increases and average daily opioid amount (mg equivalents of morphine). Secondary objectives include Weight, Appetite, N/V, O2 Saturation, Self-reported data points from the modified Edmonton Assessment Scale.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Alert adults
* requiring opioids for pain management (routine)
* cancer diagnosis or non-cancer diagnosis as their terminal illness

Exclusion Criteria:

* pregnant women
* Age < 18
* minimally or unresponsive patients unable to take oral medications
* agitated combative patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Zanker, MD, Principal Investigator — The Connecticut Hospice Inc.
Locations (1):
- The Connecticut Hospice Inc., Branford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment of Terminal Patients with pain and receiving routine opioid therapy within an inpatient Hospice Hospital setting commencing 05/10/2017 and ending 8/5/2022
Pre-assignment Details: Participants were excluded from participating if they were unable to take orally administered medications.
Period: Overall Study
Arm/Group | Single Treatment Arm
Started | 66
Completed | 58
Not Completed | 8
Not completed — Adverse Event | 2
Not completed — Less Than 3 Days of Data | 6

BASELINE CHARACTERISTICS:
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 66
Age, Categorical [Count of Participants; unit: Participants] — Age in years at time of study enrollment
  Participants
    <=18 years | 0
    Between 18 and 65 years | 26
    >=65 years | 40
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [60.25 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 64
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 60
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 66
Diagnosis Category [Count of Participants; unit: Participants]
  Cancer | 55
  Non-Cancer | 11

OUTCOME MEASURES:

1. Primary Outcome: Primary Reduction of Pain
Description: A numeric pain scale (Units on a scale with the higher number indicating worse pain) was used to assess pain from a range of 0 to 10.
Time Frame: minumum 3 days
Population: Patients in hospice care on regular scheduled opioid administration for pain management.
Measure: Mean (Standard Deviation); unit: units on a scale from 0 to 10
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 66
units on a scale from 0 to 10
  Pain level at baseline | 2.55 (2.46)
  Pain level on the last day of study | 1.40 (2.17)

2. Primary Outcome: Reduction in Overall Opioid Utilization
Description: Reduction in overall opioid utilization was measured in units of mg after converting every patient's opioids into equivalent doses (e.g. 2mg of oral dilaudid = 1/4 oral morphine), with a stabilization or reduction in Morphine Mg Equivalents indicating a positive result.
Time Frame: minimum of 3 days
Measure: Mean (Standard Deviation); unit: medical morphine equivalents (mg)
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 66
medical morphine equivalents (mg)
  Opiates administered at Baseline | 309.84 (775.62)
  Opiates administered at the end of study | 285.54 (430.76)

3. Secondary Outcome: Improvement in Overall Patient Well Being
Description: A modified Edmonton Assessment Scale was used. The Edmonton Symptom Assessment System (ESAS) is a questionnaire used to rate the intensity of common symptoms experienced by cancer patients, including pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, well-being, and shortness of breath. A scale of 1 to 10 was used, where, 1 corresponds to the best well-being and 10 corresponds to the worst well-being.
Time Frame: minimum 3 days
Measure: Mean (Standard Deviation); unit: score on a scale from 1 to 10
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 66
score on a scale from 1 to 10
  Overall well-being at Baseline | 3.31 (2.64)
  Overall well-being at the end of study | 2.42 (2.73)

4. Secondary Outcome: Weight Stabilization With Increased Appetite
Description: A modified Edmonton Assessment Scale was used. The Edmonton Symptom Assessment System (ESAS) is a questionnaire used to rate the intensity of common symptoms experienced by cancer patients, including pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, well-being, and shortness of breath.
  Appetite was analyzed as an ordinal variable where 1 = finished 0~25% of meal, 2 = 25~50% of meal, 3 = 50~75% of meal, 4 = 75~100% of meal.
Time Frame: minimum 3 days
Measure: Mean (Standard Deviation); unit: units on a scale from 1 to 4
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 66
units on a scale from 1 to 4
  Appetite at Baseline | 1.93 (1.01)
  Appetite at the end of study | 1.70 (1.07)

5. Secondary Outcome: Improved Oxygen Saturation
Description: Oxygen saturation was reported as a percentage, the greater the % O2 saturation the more positive the outcome.
Time Frame: minimum 3 days
Measure: Mean (Standard Deviation); unit: percent
Groups:
- Single Treatment Arm: Marijuana adjuvant treatment group utilizing scheduled opioid therapy in inpatient hospice hospital setting Medical Marijuana: oral capsule, high ratio CBD:THC
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 66
percent
  O2 Saturation at Baseline | 94.86 (2.53)
  O2 Saturation at the end of study | 94.10 (2.55)

6. Secondary Outcome: Reduction or Prevention of Nausea and Vomiting
Description: A modified Edmonton Assessment Scale was used; the scale is a numeric 0-10 scale (Units on a scale where the higher the number the more nausea and vomiting the patient experienced).
Time Frame: minimum 3 days
Measure: Mean (Standard Deviation); unit: units on a scale from 0 to 10
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 66
units on a scale from 0 to 10
  Nausea at Baseline | 0.46 (1.33)
  Nausea at the end of study | 0.17 (0.74)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the entire duration for which each patient was enrolled in the study (minimum of 3 days).
Description: The definitions of adverse event and serious adverse event do not differ from the definitions provided by clinicaltrials.gov.
  Adverse event data was collected by inpatient-care nursing staff members who continuously monitored each patient throughout their time enrolled in the study.
Groups:
- Medical Marijuana Treatment Arm: Because this is a single-arm study, all 66 patients included in the study were in the treatment arm, and were administered medical marijuana. All 66 patients were in hospice care and were followed up until either 1) death or 2) unable to take the medication by mouth anymore. Therefore, the study was expected to have 100% all-cause mortality.
Arm/Group | Medical Marijuana Treatment Arm
All-Cause Mortality (participants affected / at risk) | 66/66
Serious Adverse Events (participants affected / at risk) | 1/66
Other Adverse Events (participants affected / at risk) | 1/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Medical Marijuana Treatment Arm (N=66)
Panic Attack (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Medical Marijuana Treatment Arm (N=66)
Dizziness (General disorders) | 1

LIMITATIONS AND CAVEATS:
1. This is a single-arm study with only an intervention arm and no control. As a result, it is not possible to draw any causal conclusions. Follow-up studies are needed to further validate the preliminary signals and patterns observed in this study.
2. There were three patients who experienced a dose change in marijuana from 40mg to 80mg CBD.
3. Some outcome measurements were missing due to the inability of patients to respond to questions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-10-21): https://cdn.clinicaltrials.gov/large-docs/33/NCT03233633/Prot_SAP_000.pdf
  • Informed Consent Form (2016-10-21): https://cdn.clinicaltrials.gov/large-docs/33/NCT03233633/ICF_001.pdf